CLINICAL TRIAL: NCT04058249
Title: Accelerated Theta Burst Stimulation for Inpatients With Bipolar Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Bora Kim, Post-Doctoral Scholar, Stanford University, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 52635
Record Dates: First submitted 2019-08-05; First posted 2019-08-15 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: Bipolar Disorder, Manic; Bipolar Disorder I
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Right DLPFC aiTBS stimulation (Experimental)
  Interventions: Device: Accelerated intermittent theta-burst stimulation over right DLPFC

INTERVENTIONS:
Device: Accelerated intermittent theta-burst stimulation over right DLPFC — All participants will receive accelerated intermittent theta-burst stimulation to the right DLPFC. Stimulation intensity will be standardized at 90% of resting motor threshold adjust to the skull to cortical surface distance.
  Stimulation will be delivered to right-DLPFC using the Brainsway stimulator.

SUMMARY:
This study evaluates the efficacy of an accelerated schedule of theta-burst stimulation for treating manic episodes in bipolar disorder. In this open-label study, all participants will receive accelerated theta-burst stimulation.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established technology as therapy for treatment-resistant depression. The approved method for treatment is 10Hz stimulation for 40 minutes over the left dorsolateral prefrontal cortex (L-DLPFC). This methodology has been very successful in real-world situations. The limitations of this approach include the duration of the treatment (approximately 40 minutes per treatment session over 4-6 weeks). Recently, researchers have modified the treatment parameters to reduce treatment times with some preliminary success. In a recent study, an accelerated paradigm showed a significant antidepressant effect (90% remission rate) in individuals with treatment-resistant depression (TRD), in only 5 days. Additionally, 5 participants from this study carried a bipolar diagnosis and responded similarly, with no adverse events experienced or manic/hypomanic conversion observed during the treatment series. In parallel to this, evidence in the literature shows that right prefrontal rapid TMS is safe and efficacious in the treatment of bipolar mania showing laterality opposed to the proposed effect of rapid TMS in depression.

The current trial intends to utilise this modified design, i.e., an accelerated theta burst stimulation treatment over the right prefrontal cortex, for manic episodes in bipolar disorder. The trial also aims to look at the change in clinical measures and neuroimaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between the ages of 18 and 80 years at the time of screening.
* Able to read, understand, and provide written, dated informed consent prior to screening. Proficiency in English sufficient to complete questions and follow instructions during fMRI assessments and aiTBS interventions
* Stated willingness to adhere to all study procedures, including availability for the duration of the study, and to communicate with study personnel about adverse events and other clinically important information
* Primary diagnosis of Bipolar I or II Disorder according to the Diagnosis and Statistical Manual of Mental Disorders, 5th edition (DSM-5)
* Currently experiencing a hypomanic or manic episode according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, 5th edition (DSM-5)
* YMRS score of ≥12 at screening.
* Access to ongoing psychiatric care after completion of the study.
* Must be adherent or agreeable to pharmacotherapy per clinical standard of care at screening.
* Patients who are in both voluntary and involuntary hold.
* In good general health, as evidenced by medical history.
* For females of reproductive potential: use of highly effective contraception.

Exclusion Criteria:

* Currently pregnant or breastfeeding.
* Primary psychiatric condition other than Bipolar I or II Disorder requiring treatment other than stable comorbid anxiety disorder.
* Diagnosis of Intellectual Disability or Autism Spectrum Disorder
* Current moderate or severe substance use disorder or demonstrating signs of acute substance intoxication or withdrawal
* Active suicidal ideation (defined as an M-SSI > 8)
* History of significant neurologic disease, including dementia, Parkinson's or Huntington's disease, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma
* Contraindication to receiving rTMS (e.g., metal in head, history of seizure, known brain lesion)
* Contraindication to MRI (e.g. ferromagnetic metal in their body)
* Treatment with another investigational drug or other intervention within the study period
* Any other condition deemed by the PI to interfere with the study or increase risk to the participant
* Current unmanageable psychosis that the PI believes would interfere with treatment
* Any history of psychosurgery
* Depth-adjusted aiTBS treatment dose > 65% maximum stimulator output (MSO).
* Any other condition deemed by the PI to interfere with the study or increase risk to the participant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Batail, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Right DLPFC aiTBS Stimulation: Accelerated intermittent theta-burst stimulation over right DLPFC. Stimulation intensity standardized at 90% of resting motor threshold adjust to the skull to cortical surface distance.
Period: Overall Study
Arm/Group | Right DLPFC aiTBS Stimulation
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Right DLPFC aiTBS Stimulation
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Time Frame: 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Right DLPFC aiTBS Stimulation
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Young Mania Rating Scale [YMRS] Score
Description: The Y-MRS is an 11-item clinician-rated instrument for assessing the severity of manic episodes. A severity rating is assigned to each of the 11 items (Elevated mood, Increased motor activity-energy, Sexual interest, Sleep, Irritability, Speech, Language-thought disorder, Thought content, Disruptive-aggressive behavior, Appearance, Insight), based on the participant's subjective report of his or her condition over the previous 48 hours and the clinician's observations during the interview, with the emphasis on the latter. Seven of the 11 items are rated on a scale of 0-4 and 4 of the items are rated on a scale of 0-8, with higher scores indicating greater severity of symptoms. The Y-MRS total score for each participant is the sum of the ratings for the 11 individual items, and can range from 0-60, with higher scores indicating greater severity of symptoms.
Time Frame: Baseline, day 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Right DLPFC aiTBS Stimulation
Number analyzed (Participants) | 1
score on a scale
  Baseline | 15 (NA) — Standard deviation not calculable for n of 1
  Day 6 | 0 (NA) — Standard deviation not calculable for n of 1

ADVERSE EVENTS:
Time Frame: 6 days
Arm/Group | Right DLPFC aiTBS Stimulation
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT04058249/Prot_SAP_000.pdf